CLINICAL TRIAL: NCT07208903
Title: Psychological Evaluation of the Parental Experience of Newborn Screening for Infantile Spinal Muscular Atrophy in the Grand Est and Nouvelle-Aquitaine Regions
Acronym: PSYSMA
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9759
Record Dates: First submitted 2025-09-23; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Spinal Muscular Atrophy (SMA); Spinal Muscular Atrophy Type I
MeSH Terms: conditions — Muscular Atrophy, Spinal; Spinal Muscular Atrophies of Childhood | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Treated positive screening group: Parents of children with a positive neonatal genetic screening result who received treatment (<4 SMN2 copies)
  Interventions: Behavioral: focus group discussions
- Untreated positive screening group: Parents of children with a positive neonatal genetic screening result who did not receive treatment (≥4 SMN2 copies)
  Interventions: Behavioral: focus group discussions
- False-negative screening group: Parents of children with a false-negative neonatal genetic screening result (diagnosed secondarily)
  Interventions: Behavioral: Interview with the psychologist

INTERVENTIONS:
Behavioral: focus group discussions — These sessions will address:
  * emotional reactions to the disclosure of the result
  * perceptions and representations of the disease and its treatment
  * the impact on the parent-child relationship
  * the lived experience of neonatal screening and the perception of the support provided
  Groups: Treated positive screening group; Untreated positive screening group
Behavioral: Interview with the psychologist — These sessions will address:
  * emotional reactions to the disclosure of the result
  * perceptions and representations of the disease and its treatment
  * the impact on the parent-child relationship
  * the lived experience of neonatal screening and the perception of the support provided
  Groups: False-negative screening group

SUMMARY:
The systematic inclusion of spinal muscular atrophy (SMA) in France's neonatal genetic screening (NGS) program, scheduled for September 2025, represents a major milestone in public health. While this screening enables early detection and therapeutic intervention before symptom onset, it also raises psychological and ethical challenges that remain underexplored-particularly during the highly sensitive postpartum period.

Currently, data on parental experiences following a positive SMA NGS result are scarce, fragmented, and largely derived from North American studies or from metabolic screening contexts. Early publications highlight high levels of parental anxiety, dissatisfaction with the quality of result disclosure, and difficulties in processing complex medical information in a short, emotionally charged timeframe. These findings underscore the need for a deeper understanding of the subjective processes at play in this situation.

The PSYSMA project is designed as an ancillary study to the DEPISMA trial. Its aim is to retrospectively explore parents' lived experiences, their psychosocial support needs, and the impact of NGS on family dynamics and the parent-child relationship. Special attention is given to cases with uncertain results (e.g., ≥4 SMN2 copies without treatment) and false negatives, which remain poorly documented but may trigger unique forms of parental anxiety or adaptation.

This research is justified by two main needs:

* to guide public health policy toward integrating psychological support from the earliest stages of screening, in line with French National Health Authority (HAS) recommendations;
* to generate new knowledge transferable to other genetic diseases that may be included in future neonatal screening programs.

The overarching goal is to retrospectively investigate the psychological experience of parents confronted with a positive or false-negative SMA NGS result, in order to analyze its subjective, emotional, and relational effects, as well as related needs for psychological support.

Study objectives :

* Compare parental experiences according to the nature of the result (with or without treatment indication).
* Identify psychosocial support needs, including for siblings.
* Assess anxiety, depression, and post-traumatic symptoms associated with NGS.
* Explore the broader impact on family functioning, particularly in relation to genetic counseling and communication within the extended family.

ELIGIBILITY:
Inclusion Criteria:

* Be the parent of a child included in the DEPISMA study, born in the Grand Est or Nouvelle-Aquitaine region;
* Have received a positive or false-negative result from the neonatal SMA screening;
* Be an adult at the time of inclusion;
* Be proficient in French in order to participate in a focus group or an individual interview, and to complete the self-administered questionnaires;
* Have been informed of the NNS result for at least 4 months, to allow sufficient time for a subjective reflection

Exclusion Criteria:

* Parent who is not sufficiently proficient in French to participate in focus groups or complete questionnaires
* Death of the child who was screened

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study participants are parents of children born in the Grand Est or Nouvelle-Aquitaine regions who received a positive or false-negative result from the neonatal screening for SMA during DEPISMA study. They must be adults who are proficient in French and have had at least four months to process the screening results.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2025-10-20 (Estimated); Primary Completion 2026-10-20 (Estimated); Study Completion 2026-10-20 (Estimated)

PRIMARY OUTCOMES:
Quantitative: Content of the questionnaires completed at the inclusion visit | Month 4, plus or minus 2 months
  Scores on the IES-R scale (Impact of Event Scale) for post-traumatic stress. Minimum value: 0 (if the person selects "not at all" for all 22 items).
  Maximum value: 88 (if the person selects "extremely" for all 22 items). Interpretation: Higher scores reflect worse outcomes, meaning more severe post-traumatic stress symptoms (intrusion, avoidance, hyperarousal).
Qualitative: Content of interviews/focus groups at the follow-up visit regarding | Month 4, plus or minus 2 months
  Emotional reactions to the announcement Representations of the illness and its treatment Impact on the parent-child relationship Experience of the screening process and the perception of support received
Quantitative: Content of the questionnaires completed at the inclusion visit | Month 4, plus or minus 2 months
  Scores on the HADS scale (Hospital Anxiety and Depression Scale) for anxiety symptoms.
  Structure: 14 items total, split into two subscales:
  * HADS-A (Anxiety) - 7 items
  * HADS-D (Depression) - 7 items Minimum value: 0 (no symptoms). Maximum value: 21 per subscale (if all items scored at the maximum of 3). but 42 total if both subscales are summed. Interpretation: Higher scores reflect a worse outcome, meaning greater anxiety and/or depressive symptom severity.

IPD SHARING:
Plan to Share IPD: No